CLINICAL TRIAL: NCT05429580
Title: Efficacy of Prophylactic Tranexamic Acid Use After Vaginal Delivery According to Postpartum Hemorrhage Risk: Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Prophylactic Tranexamic Acid Use After Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-KAEK-25 2021/07-22
Record Dates: First submitted 2022-06-18; First posted 2022-06-23 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Postpartum Hemorrhage; Vaginal Delivery; Prophylactic Tranexamic Acid Use
Keywords: tranexamic acid; vaginal delivery; postpartum hemorrhage; active management of vaginal delivery
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Glucose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postpartum bleeding risks as low-risk (Other): The patients were divided into two groups according to their postpartum bleeding risks as low-risk (240 patients) and high-risk (240 patients), and then the patients in each group were randomly divided into two groups, and some of these pregnant women were given intravenous tranexamic acid and some were given placebo.
  Interventions: Drug: Tranexamic acid; Other: 5% Dextrose
- postpartum bleeding risks as high-risk (Other): The patients were divided into two groups according to their postpartum bleeding risks as low-risk (240 patients) and high-risk (240 patients), and then the patients in each group were randomly divided into two groups, and some of these pregnant women were given intravenous tranexamic acid and some were given placebo.
  Interventions: Drug: Tranexamic acid; Other: 5% Dextrose

INTERVENTIONS:
Drug: Tranexamic acid — given intravenous tranexamic acid
Other: 5% Dextrose — given placebo.

SUMMARY:
In this study, our aim was to evaluate the effectiveness of prophylactic tranexamic acid use after vaginal delivery in pregnant women aged 18-45 years and 34-42 weeks according to the risk of postpartum hemorrhage.

DETAILED DESCRIPTION:
It was carried out as a double-blind prospective randomized controlled Phase 4 drug study with 480 singleton pregnant women in Bursa Yüksek İhtisas Training and Research Hospital between September 1, 2021 and February 28, 2022. The patients were divided into two groups as low risk (240 patients) and high risk (240 patients) according to their postpartum hemorrhage risks, and the patients in each group were randomly divided into two groups. Group 1: were given intravenous tranexamic acid and group 2: were given placebo. The blood loss at the 3rd and 4th stages of labor was calculated by weighing the blood collected with the help of a collecting pochette and using the estimated blood loss formula.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women
* woman between the ages of 18-45 years
* woman who gave birth at 34 weeks and above

Exclusion Criteria:

* Pregnancies with less than 1 hour period between hospitalization and delivery
* Women with placenta previa, invasion anomaly or diagnosis of abruptio placentae
* Women with previous uterine surgery or cesarean section
* Women with a history of thromboembolism
* women with serious illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The loss of blood at the 3rd and 4th stages of labor | 6 month
  It was calculated by weighing the blood collected with the help of collecting bag and using the estimated blood loss formula.

SECONDARY OUTCOMES:
The success of tranexamic acid in patients grouped according to the postpartum bleeding risk scale | 6 months
  The success of tranexamic acid in patients grouped according to the postpartum bleeding risk scale association with atony, need for blood transfusion, need for extra uterotonics, and the gastrointestinal side effects of tranexamic acid such as nausea, vomiting, and diarrhea were evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)